CLINICAL TRIAL: NCT06063590
Title: An Open-Label Single-Arm Phase I/IIa Study to Evaluate the Safety of Human Allogenic Bone-Marrow-Derived Mesenchymal Stromal Cell Product StromaForte in Patients With Aging Frailty
Brief Title: A Study to Evaluate Allogenic Bone-Marrow Mesenchymal Stromal Cell Product StromaForte in Aging Frailty Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cellcolabs Clinical SPV Limited (Industry)
Collaborators: PDC-CRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-Frailty Study-2022
Record Dates: First submitted 2023-08-30; First posted 2023-10-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Aging Frailty

STUDY DESIGN:
Intervention Model Description: The patients will be assigned into one group receiving allogeneic bone marrow (BM)- derived Mesenchymal Stromal Cell (MSC) formulated in infusion solution (sodium chloride supplemented with human serum albumin Pre-screening visit will be conducted within 7 days of the screening visit then eligible patient will participate in the Study for approximately 6 months and will have a total of 5 on-site visits, including a screening visit, a treatment administration visit, and 3 follow-up visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC arm (Experimental): The patients will be receiving allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cell (MSC) formulated in infusion solution (sodium chloride supplemented with human serum albumin) in a low intravenous infusion of 100 millions MSCs within approximately 30 min
  Interventions: Biological: StromaForte

INTERVENTIONS:
Biological: StromaForte — 100 millions allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cell (MSC) formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion in approximately 30 min

SUMMARY:
This phase I/IIa study in frail patients is designed to assess the safety of intravenous human allogenic bone marrow-derived mesenchymal stromal cell product StromaForte by reporting the number of adverse events assessed by Common Terminology Criteria. 12 male and female patients aged 60 to 85 years will be enrolled.

DETAILED DESCRIPTION:
Frailty is theoretically defined as a clinically recognizable state of increased vulnerability resulting from aging-associated decline in reserve and function across multiple physiologic systems such that the ability to cope with every day or acute stressors is comprised. In the absence of a gold standard, frailty has been operationally defined by Fried et al. as meeting three out of five phenotypic criteria indicating compromised energetics: low grip strength, low energy, slowed waking speed, low physical activity, and/or unintentional weight loss.

One major factor proposed to contribute to frailty and related epigenetic dysregulation is stem cell loss. In order to treat this multifactorial dysregulation, stem cell therapy is an interesting strategy, and MSCs are a particularly tempting candidate. MSCs are an immune-privileged somatic progenitor cell type that is multipotent, self-renewing, and relatively simple to harvest (bone marrow harvest), isolate, and grow. MSCs are proven to regulate the body's immune response in many diseases and exert anti-inflammatory effects.

Following their discovery over 50 years ago, mesenchymal stromal cells (MSCs) have become one of the most studied cellular therapeutic products by both academia and industry due to their regenerative potential and immunomodulatory properties. The promise of MSCs as a therapeutic modality has been demonstrated in a number of preclinical studies as well as in clinical setting. Stromaforte cells which will be used in this study is developed within CELLCOLABS AB which is a parent company to Cellcolabs Clinical SPV Limited and were generated following the same protocol established over the last 20 years by scientists CELLCOLABS AB at the Karolinska Institute in Sweden.

Currently completed in vivo studies on rats, rabbits and mice models showed that MSCs could attenuate sarcopenia via increasing skeletal muscle weight and myofiber cross-sectional area. The physical performance including muscle strength as well as endurance were significantly enhanced. In addition, MSCs have capability to activate resident skeletal muscle stem cells, which lead to myogenesis and differentiation of muscle tissues. The positive results provide novel insights into sarcopenia intervention, suggesting a potential role for MSC therapy in aging frailty. This study which has been designed to evaluate the safety of intravenous human allogenic bone marrow-derived mesenchymal stromal cell product StromaForte in frail patients before further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and comply with all procedures required by the protocol
* Aged ≥ 60 and ≤ 85 years at the time of signing the informed consent form,
* Have a Canadian Study on Health and Aging (CSHA) Clinical Frailty Scale score of 5 "mildly frail" or 6 "moderately frail"
* Have a 6-minute walk distance of > 200m and < 400 m
* Have a serum TNF-alpha level ≥2.5 pg/ml

Exclusion Criteria:

* Unwilling or unable to perform any of the assessments required by the protocol
* Have a diagnosis of any disabling neurologic disorder, including, but not limited to, Parkinson's disease, Amyotrophic Lateral Sclerosis, multiple sclerosis, cerebrovascular accident with residual deficits (e.g., muscle weakness or gait disorder), or diagnosis of dementia
* Have a score of 24 or lower on the Mini Mental State Examination (MMSE)
* Have poorly controlled blood glucose levels (HbA1c >8.0%)
* Have a clinical history of malignancy within 2.5 years (i.e., patients with prior malignancy must be cancer free for 2.5 years) except curatively treated basal cell carcinoma, melanoma in situ or cervical carcinoma
* Have any condition that limits lifespan to < 1 year according to the Principal Investigator discretion
* Have autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus)
* Undergoes chronic immunosuppressant therapy such as high-dose corticosteroids or TNF-α antagonists (prednisone use at doses of < 5 mg daily is allowed)
* Hepatitis B virus positive
* Viraemic Hepatitis C virus, HIV-1/2 or syphilis positive
* Have a resting blood oxygen saturation of <93% (measured by pulse oximetry)
* Known or suspected alcohol or drug abuse within three years preceding Screening
* Have a known hypersensitivity to dimethyl sulfoxide (DMSO)
* An organ transplant recipient (other than transplantation for corneal)
* Actively listed (or expected future listing) for transplant of any organ (other than corneal transplant)
* Have any clinically important abnormal screening laboratory values, including, but not limited to: i. Haemoglobin <10.0 g/dL, ii. White blood cell <2,500/ul, or platelet count <100,000/ul iii. Liver dysfunction evidenced by enzymes (AST and ALT) > 3 times the upper limit of normal (ULN)
* Coagulopathy with international normalized ratio (INR) >1.3 not due to a reversible cause (e.g., warfarin and/or Factor Xa inhibitors)
* Uncontrolled hypertension (resting systolic blood pressure >180 mm Hg or diastolic blood pressure of > 110 mm Hg at Screening)
* Have unstable angina pectoris, uncontrolled or severe peripheral artery disease within the previous 3 months
* Have congestive heart failure defined by New York Heart Association (NYHA) Class III or IV, or an ejection fraction of <25
* Have a coronary artery bypass surgery, angioplasty, or peripheral vascular disease revascularization or a myocardial infarction within previous 3 months
* Have severe pulmonary dysfunction: acute exacerbation of chronic obstructive lung disease stage III or IV (Gold classification), and/or PaO2 levels <60 mmHg
* Have a partial ileal gastric bypass, or other significant intestinal malabsorption
* Have advanced liver or renal disease
* Have cognitive or language barriers that prohibit obtaining informed consent or any study elements
* (or participated within the previous 30 days of consent) in an investigational Currently hospitalized or living in an assisted living facility or a long-term care facility
* Currently participating therapeutic or device trial
* Have a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the patient's participation for the full duration of the study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-28 (Estimated); Primary Completion 2024-11-28 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 days post-infusion
  To assess the safety and tolerability after 28 days of injection by reporting the number of adverse events assessed by Common Terminology Criteria For Adverse Events (CTCAE) which is the Incidence of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities determined per the Investigator's judgment along with others Adverse Events and Serious Adverse events

SECONDARY OUTCOMES:
Change in TNF-alpha | From baseline to 6 months
  Change in tumor necrosis factor α TNF-α from baseline to 6 months (baseline to 28-, 84-, and 168-days post-infusion.)
Change in C Reactive Protein (CRP) | From baseline to 6 months
  Change in C Reactive Protein (CRP) from baseline to 6 months (baseline to 28-, 84-, and 168-days post-infusion.)
Change in Interleukin-6 (IL-6) | From baseline to 6 months
  Change in Interleukin-6 (IL-6) from baseline to 6 months (baseline to 28-, 84-, and 168-days post-infusion.)
Change in Complete Blood Count (CBC) in peripheral blood with differential | From baseline to 6 months
  Change in Complete Blood Count (CBC) in peripheral blood with differential from baseline to 6 months (baseline to 28-, 84-, and 168-days post-infusion.)

OTHER OUTCOMES:
Change in the 6-minute walk test | From baseline to 6 months
  Change in the 6-minute walk test (6-MWT) from baseline to 28-, 84- and 168- days post infusion.
Change in hand grip strength | From baseline to 6 months
  Change in hand grip strength (dynamometry) from baseline to 28 ,84 and 168 days post-infusion.
Change in EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS) | From baseline to 6 months
  Change in EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS) from baseline to 84-, and 168-days post-infusion. The maximum score of EQ-5D is 1 which indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
Change in Multidimensional Fatigue Inventory (MFI) | From baseline to 6 months
  Change in Multidimensional Fatigue Inventory (MFI) from baseline to 84-, and 168-days post-infusion. MFI-20 has an even proportion of positively and negatively worded items that are rated on a 5-point Likert scale. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores.
Change in 36-Item Short Form health survey (SF-36) | From baseline to 6 months
  Change in 36-Item Short Form health survey (SF-36) from baseline to 84-, and 168-days post-infusion. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Change in the MMSE | From baseline to 6 months
  Change in the Mini Mental State Examination (MMSE) criteria after 6 months. The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Fahti Yousef, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Burjeel Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No